CLINICAL TRIAL: NCT06273540
Title: Phase 1, Double-Blind, Placebo-Controlled, Parallel Group Study to Assess Potential Interactions Between Intravenous Cocaine and Oral STP7
Brief Title: Phase1, STP7 Cocaine Drug-Drug Interaction Study
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Stalicla SA (Industry)
Collaborators: National Institute on Drug Abuse (NIDA) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: STA-P7-C001; C-043-2023 (Other Grant/Funding Number: NIDA)
Record Dates: First submitted 2024-01-04; First posted 2024-02-22 (Actual); Last update posted 2025-12-02 (Actual); Status verified 2025-10

CONDITIONS: Cocaine Use Disorder
Keywords: STP7; mavoglurant; Cocaine; AFQ056; metabotropic glutamate receptor 5; mGluR5; CUD
MeSH Terms: interventions — mavoglurant; Cocaine

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- STP7 (mavoglurant) modified release film-coated tablet (Experimental): Participants will take STP7 (mavoglurant) twice a day (BID) from Days 3 to 9 according to the following dosing schedule:
  * Day 3: 50 mg BID;
  * Day 4: 100 mg BID;
  * Days 5-9: 200 mg BID,
  * Day 10: 200 mg only the morning dose.
  Morning STP7 (mavoglurant) doses must be taken within 30 minutes of beginning a meal.
  Interventions: Drug: STP7 (mavoglurant)
- Placebo (Placebo Comparator): Participants will take matched placebo twice a day (BID) from Days 3 to 9 and only the morning dose on Day 10.
  Morning Placebo must be taken within 30 minutes of beginning a meal.
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: STP7 (mavoglurant) — STP7 (mavoglurant) twice a day (BID) from Days 3 to 9 according to the following dosing schedule: Day 3: 50 mg BID; Day 4: 100 mg BID; Days 5-9: 200 mg BID, and will take only the morning dose of STP7 (200 mg) on Day 10.
  Cocaine / Saline
  Participants will undergo cocaine/saline i.v. challenge sessions according to the schedule and doses:
  * Screening (Session 1, Day -2): 20 mg cocaine, followed by a saline infusion, followed by 40 mg cocaine
  * Baseline (Session 2, Day 1): saline or 20 mg cocaine followed by either 20 mg cocaine or saline.
  * Baseline (Session 3, Day 2): saline or 40 mg cocaine followed by either 40 mg cocaine or saline.
  * Treatment (Session 4, Day 9): saline or 20 mg cocaine followed by either 20 mg cocaine or saline.
  * Treatment (Session 5, Day 10): saline or 40 mg cocaine followed by either 40 mg cocaine or saline.
  Other Names: Cocaine; Saline infusion
  Arms: STP7 (mavoglurant) modified release film-coated tablet
Drug: Placebo — Placebo twice a day (BID) from Days 3 to 9 BID, and will take only the morning dose of Placebo on Day 10.
  Cocaine / Saline
  Participants will undergo cocaine/saline i.v. challenge sessions according to the schedule and doses:
  * Screening (Session 1, Day -2): 20 mg cocaine, followed by a saline infusion, followed by 40 mg cocaine
  * Baseline (Session 2, Day 1): saline or 20 mg cocaine followed by either 20 mg cocaine or saline.
  * Baseline (Session 3, Day 2): saline or 40 mg cocaine followed by either 40 mg cocaine or saline.
  * Treatment (Session 4, Day 9): saline or 20 mg cocaine followed by either 20 mg cocaine or saline.
  * Treatment (Session 5, Day 10): saline or 40 mg cocaine followed by either 40 mg cocaine or saline.
  Other Names: Cocaine; Saline infusion
  Arms: Placebo

SUMMARY:
This is a double-blind, placebo-controlled, parallel group study to compare the effects of STP7 (mavoglurant) vs placebo control on i.v. cocaine's physiological and subjective effects in non-treatment seeking, cocaine-experienced males or females participants between 18 and 59 years of age.

The primary objective of this study is to determine if there are clinically meaningful interactions between oral STP7 (mavoglurant) treatment concurrent with 20 and 40 mg i.v. cocaine infusions by measuring adverse events and cardiovascular responses including heart rate, blood pressure, and electrocardiogram (including corrected QT interval).

The secondary objectives are:

* To evaluate whether administration of STP7 (mavoglurant) alters the pharmacokinetics of cocaine and/or its major metabolite, benzoylecgonine.
* To determine the pharmacokinetic of STP7 (mavoglurant) administered at a dose of 200 mg twice a day.
* To evaluate whether STP7 (mavoglurant) treatment alters the subjective effects of cocaine measured by Visual Analog Scales (VAS) and Brief Substance Craving Scale (BSCS).

ELIGIBILITY:
Inclusion Criteria:

1. Be participants who are cocaine-experienced and not seeking treatment for cocaine use disorder.
2. Males and females between 18 and 59 years of age, inclusive.
3. Have a body mass index (BMI) within a range of 17.0 to 36.0 kg/m2 and a minimum weight of at least 50.0 kg at screening.
4. Have experience using cocaine by the smoked or i.v. route at least 6 times in the past 12 months prior to clinic intake (Day -3) and at least one use (smoked, i.v., or nasal route) within the past 3 months.
5. Provide a urine sample positive for cocaine at least once during screening (Days -28 to -4).
6. Be able to verbalize understanding of consent form, able to provide written informed consent, and verbalize willingness to complete study procedures.
7. A female study participant must meet one of the following criteria:

   If of childbearing potential - agrees to use one of the accepted contraceptive regimens from at least 30 days prior to the first administration of the study medication, during the study, and for at least 30 days after the last dose of the study medication. An acceptable method of contraception includes one of the following:

   i. Abstinence from heterosexual intercourse ii. Hormonal contraceptives (injectable/implant/insertable hormonal birth control products, transdermal patch) iii. Intrauterine device (with or without hormones) OR agrees to use a double barrier method (e.g. condom and spermicide) during the study and for at least 30 days after the last dose of the study medication. If a female of non-childbearing potential - should be surgically sterile (i.e. has undergone complete hysterectomy, bilateral oophorectomy, or tubal ligation/occlusion) or in a menopausal state (at least 1 year without menses), as confirmed by FSH levels.

   A male study participant that engages in sexual activity that has the risk of pregnancy must agree to use a double barrier method (e.g. condom and spermicide) and agree to not donate sperm during the study and for at least 90 days after the last dose of the study medication.
8. Be able to comply with protocol requirements, rules and regulations of the study site, and be likely to complete all the study treatments.

Exclusion Criteria:

1. Have a current or past history of seizure disorder, including alcohol- or stimulant-related seizure, febrile seizure, or significant family history of idiopathic seizure disorder.
2. Have any previous medically adverse reaction to cocaine, including loss of consciousness, chest pain, paranoid reaction or seizure.
3. Have clinically significant findings in the opinion of an investigator based on the MINI (version 7.0) neuropsychiatric interview.
4. Be pregnant or lactating.
5. Have a sitting systolic blood pressure > 140 mmHg, diastolic blood pressure > 90 mmHg and heart rate > 100 beats per minute at screening and clinic intake.
6. Have a history of liver disease or current elevation of liver function test (LFT) values as follows:

   * aspartate aminotransferase (AST) >2x the upper limit of normal
   * alanine aminotransferase (ALT) >2 × the upper limit of normal.
7. Have a history of renal disease or current renal function test values as follows:

   * blood urea nitrogen (BUN) >2× ULN, or
   * creatinine >1.5 mg/dL.
8. Blood donation (excluding plasma donation) of approximately 500 mL within 56 days prior to screening.
9. Plasma donation within 7 days prior to screening.
10. Treatment with an investigational drug within 30 days or 5 times the half-life (whichever is longer) prior to screening.
11. Have consumed grapefruit or other foods that inhibit or induce CYP3A4 within 7 days of Study Day 1.
12. Have any clinically significant finding on medical history, physical examination, clinical laboratory test, vital signs or ECGs that contraindicate participation in the study.
13. Have a history of suicide attempts or current or recent evidence of suicidal ideation in the past 12 months based on the Columbia-Suicide Severity Rating Scale.
14. Have a positive urine drug screen upon clinic intake (Day -3) for any of the following drugs: alcohol, amphetamine/methamphetamine, barbiturates, benzodiazepines, buprenorphine, cocaine, fentanyl, 3,4 methylenedioxymethamphetamine (MDMA), methadone, phencyclidine/phenylcyclohexyl piperidine (PCP), propoxyphene, and opioids (e.g., codeine, heroin, morphine, oxycodone, etc.).
15. Have used any prescription drugs within 14 days of clinic intake or non-prescription drugs or herbal remedies within 7 days of clinic intake.
16. Be unable to distinguish between a 20 mg and 40 mg dose of cocaine i.v. based on the high effects VAS at either the 5 or 10 minute time point during the screening infusion.
17. Have a positive serology for Hepatitis B surface antigen (HBsAg), Hepatitis C antibody (HCVab), or human immunodeficiency virus (HIV).
18. Have positive results for a coronavirus disease 2019 (COVID-19) test performed after screening is complete and participant is confirmed, but prior to admission.

Ages: 18 Years to 59 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 21 (Actual)
Dates: Start 2024-04-15 (Actual); Primary Completion 2024-10-07 (Actual); Study Completion 2024-10-07 (Actual)

PRIMARY OUTCOMES:
Incidence of Treatment-Emergent Adverse Events. | On day -2, day -1, day 1, day 2, day 3, day 4, day 5, day 6, day 7, day 8, day 9, day10, day 11, day 12 and the follow-up (window from day 19 to day 26).
  Any events spontaneously reported by the participant or observed by the investigative staff will also be recorded.
Heart Rate response following the STP7 treatment with the cocaine infusion. | Collected at day -2 at the time points (relative to the first infusion of the day): -30, - 15, 5, 10, 15, 20, 25, 30, 45, 55, 65, 70, 75, 80, 85, 90, 105, 115, 125, 130, 135, 140, 145, 150, 165, 180, 210, 240, 270, 300, 330 and 360 minutes
  Change of the Heart Rate.
Heart Rate response following the STP7 treatment with the cocaine infusion. | Collected at day 1, day 2, day 9 and day 10 at the time points (relative to the first infusion of the day): -30, -15, 5, 10, 15, 20, 25, 30, 45, 55, 65, 70, 75, 80, 85, 90, 105, 120, 150, 180, 210, 240, 270 and 300 minutes
  Change of the Heart Rate.
Blood Pressure (diastolic) response following the STP7 treatment with the cocaine infusion . | Collected at day -2 at the time points (relative to the first infusion of the day): -30, - 15, 5, 10, 15, 20, 25, 30, 45, 55, 65, 70, 75, 80, 85, 90, 105, 115, 125, 130, 135, 140, 145, 150, 165, 180, 210, 240, 270, 300, 330 and 360 minutes
  Change of the diastolic Blood Pressure.
Blood Pressure (diastolic) response following the STP7 treatment with the cocaine infusion. | Collected at day 1, day 2, day 9 and day 10 at the time points (relative to the first infusion of the day): -30, -15, 5, 10, 15, 20, 25, 30, 45, 55, 65, 70, 75, 80, 85, 90, 105, 120, 150, 180, 210, 240, 270 and 300 minutes
  Change of the diastolic Blood Pressure.
Blood Pressure (systolic) response following the STP7 treatment with the cocaine infusion. | Collected at day -2 at the time points (relative to the first infusion of the day): -30, - 15, 5, 10, 15, 20, 25, 30, 45, 55, 65, 70, 75, 80, 85, 90, 105, 115, 125, 130, 135, 140, 145, 150, 165, 180, 210, 240, 270, 300, 330 and 360 minutes
  Change of the systolic Blood Pressure.
Blood Pressure (systolic) response following the STP7 treatment with the cocaine infusion. | Collected at day 1, day 2, day 9 and day 10 at the time points (relative to the first infusion of the day): -30, -15, 5, 10, 15, 20, 25, 30, 45, 55, 65, 70, 75, 80, 85, 90, 105, 120, 150, 180, 210, 240, 270 and 300 minutes
  Change of the systolic Blood Pressure.
ECG changes (HR) following the STP7 treatment with the cocaine infusion. | As collected at day -2 at -10 minutes and at 5, 10, 15, 30, 45, 65, 70, 75, 90, 105, 125, 130, 135, 150, 165, 180 and 360 minutes after the first infusion.
  Changes in ECG (HR) following STP7 treatment with the cocaine infusion at screening.
ECG changes (RR) following the STP7 treatment with the cocaine infusion. | As collected at day -2 at -10 minutes and at 5, 10, 15, 30, 45, 65, 70, 75, 90, 105, 125, 130, 135, 150, 165, 180 and 360 minutes after the first infusion.
  Changes in ECG (RR) following STP7 treatment with the cocaine infusion at screening.
ECG changes (PR) following the STP7 treatment with the cocaine infusion. | As collected at day -2 at -10 minutes and at 5, 10, 15, 30, 45, 65, 70, 75, 90, 105, 125, 130, 135, 150, 165, 180 and 360 minutes after the first infusion.
  Changes in ECG (PR) following STP7 treatment with the cocaine infusion at screening.
ECG changes (QRS) following the STP7 treatment with the cocaine infusion. | As collected at day -2 at -10 minutes and at 5, 10, 15, 30, 45, 65, 70, 75, 90, 105, 125, 130, 135, 150, 165, 180 and 360 minutes after the first infusion.
  Changes in ECG (QRS) following STP7 treatment with the cocaine infusion at screening.
ECG changes (QT) following the STP7 treatment with the cocaine infusion. | As collected at day -2 at -10 minutes and at 5, 10, 15, 30, 45, 65, 70, 75, 90, 105, 125, 130, 135, 150, 165, 180 and 360 minutes after the first infusion.
  Changes in ECG (QT) following STP7 treatment with the cocaine infusion at screening.
ECG changes (HR) following the STP7 treatment with the cocaine infusion. | As collected at day 1, day 2, day 9 and day 10 at -10 minutes and at 5, 10, 15, 30, 45, 65, 70, 75, 90, 120, 150, 180 and 300 minutes after the first infusion.
  Changes in ECG (HR) following STP7 treatment with the cocaine infusion (baseline and treatment period).
ECG changes (RR) following the STP7 treatment with the cocaine infusion. | As collected at day 1, day 2, day 9 and day 10 at -10 minutes and at 5, 10, 15, 30, 45, 65, 70, 75, 90, 120, 150, 180 and 300 minutes after the first infusion.
  Changes in ECG (RR) following STP7 treatment with the cocaine infusion (baseline and treatment period).
ECG changes (PR) following the STP7 treatment with the cocaine infusion. | As collected at day 1, day 2, day 9 and day 10 at -10 minutes and at 5, 10, 15, 30, 45, 65, 70, 75, 90, 120, 150, 180 and 300 minutes after the first infusion.
  Changes in ECG (PR) following STP7 treatment with the cocaine infusion (baseline and treatment period).
ECG changes (QRS) following the STP7 treatment with the cocaine infusion. | As collected at day 1, day 2, day 9 and day 10 at -10 minutes and at 5, 10, 15, 30, 45, 65, 70, 75, 90, 120, 150, 180 and 300 minutes after the first infusion.
  Changes in ECG (QRS) following STP7 treatment with the cocaine infusion (baseline and treatment period).
ECG changes (QT) following the STP7 treatment with the cocaine infusion. | As collected at day 1, day 2, day 9 and day 10 at -10 minutes and at 5, 10, 15, 30, 45, 65, 70, 75, 90, 120, 150, 180 and 300 minutes after the first infusion.
  Changes in ECG (QT) following STP7 treatment with the cocaine infusion (baseline and treatment period).

SECONDARY OUTCOMES:
Pharmacokinetics: Maximum Plasma Concentration [Cmax] of cocaine. | Day 2 and day 10: at 15 minutes before the first infusion, and at 5, 15, 30, 65, 75, 90, 120, 150, and 180 minutes, and at 4, 8, 12, 20 and 32 hours after the first infusion.
  Plasma concentration-time profiles of cocaine.
Pharmacokinetics: Maximum Plasma Concentration [Cmax] of benzoylecgonine. | Day 2 and day 10: at 15 minutes before the first infusion, and at 5, 15, 30, 65, 75, 90, 120, 150, and 180 minutes, and at 4, 8, 12, 20 and 32 hours after the first infusion.
  Plasma concentration-time profiles of benzoylecgonine.
Pharmacokinetics: Maximum Plasma Concentration [Cmax] of STP7. | Day 5, day 6, day 7, day 8 and day 9: prior to the morning dose and 4 hours post-dose for each day.
  Plasma concentration-time profiles of STP7.
Pharmacokinetics: Maximum Plasma Concentration [Cmax] of STP7. | Day 10, at pre-dose, 1, 2, 4, 6, 8, 12, 16, 24, 36, and 48 hours post-dose.
  Plasma concentration-time profiles of STP7.
Pharmacokinetics: time to maximum plasma concentration [Tmax] of cocaine. | Day 2 and day 10: at 15 minutes before the first infusion, and at 5, 15, 30, 65, 75, 90, 120, 150, and 180 minutes, and at 4, 8, 12, 20 and 32 hours after the first infusion.
  Time to maximum plasma concentration of cocaine.
Pharmacokinetics: time to maximum plasma concentration [Tmax] of benzoylecgonine. | Day 2 and day 10: at 15 minutes before the first infusion, and at 5, 15, 30, 65, 75, 90, 120, 150, and 180 minutes, and at 4, 8, 12, 20 and 32 hours after the first infusion.
  Time to maximum plasma concentration of benzoylecgonine.
Pharmacokinetics: time to maximum plasma concentration [Tmax] of STP7. | Day 5, day 6, day 7, day 8 and day 9: prior to the morning dose and 4 hours post-dose for each day.
  Time to maximum plasma concentration of STP7.
Pharmacokinetics: time to maximum plasma concentration [Tmax] of STP7. | Day 10, at pre-dose, 1, 2, 4, 6, 8, 12, 16, 24, 36, and 48 hours post-dose.
  Time to maximum plasma concentration of STP7.
Pharmacokinetics: area under the concentration-time curve from time 0 to time t of cocaine. | Day 2 and day 10: at 15 minutes before the first infusion, and at 5, 15, 30, 65, 75, 90, 120, 150, and 180 minutes, and at 4, 8, 12, 20 and 32 hours after the first infusion.
  Area under the concentration-time curve from time 0 to time t (AUC0-t) of cocaine.
Pharmacokinetics: area under the concentration-time curve from time 0 to time t of benzoylecgonine. | Day 2 and day 10: at 15 minutes before the first infusion, and at 5, 15, 30, 65, 75, 90, 120, 150, and 180 minutes, and at 4, 8, 12, 20 and 32 hours after the first infusion.
  Area under the concentration-time curve from time 0 to time t (AUC0-t) of benzoylecgonine.
Pharmacokinetics: area under the concentration-time curve from time 0 to time of STP7. | Day 5, day 6, day 7, day 8 and day 9: prior to the morning dose and 4 hours post-dose for each day.
  Area under the concentration-time curve from time 0 to time t (AUC0-t) of STP7.
Pharmacokinetics: area under the concentration-time curve from time 0 to time of STP7. | Day 10, at pre-dose, 1, 2, 4, 6, 8, 12, 16, 24, 36, and 48 hours post-dose.
  Area under the concentration-time curve from time 0 to time t (AUC0-t) of STP7.
Pharmacokinetics: area under the concentration-time curve from time 0 to 12 hours post-dose of cocaine. | Day 2 and day 10: at 15 minutes before the first infusion, and at 5, 15, 30, 65, 75, 90, 120, 150, and 180 minutes, and at 4, 8, 12, 20 and 32 hours after the first infusion.
  Area under the concentration-time curve from time 0 to 12 hours post-dose (AUC0-12) of cocaine.
Pharmacokinetics: area under the concentration-time curve from time 0 to 12 hours post-dose of benzoylecgonine. | Day 2 and day 10: at 15 minutes before the first infusion, and at 5, 15, 30, 65, 75, 90, 120, 150, and 180 minutes, and at 4, 8, 12, 20 and 32 hours after the first infusion.
  Area under the concentration-time curve from time 0 to 12 hours post-dose (AUC0-12) of benzoylecgonine.
Pharmacokinetics: area under the concentration-time curve from time 0 to 12 hours post-dose of STP7. | Day 5, day 6, day 7, day 8 and day 9: prior to the morning dose and 4 hours post-dose for each day.
  Area under the concentration-time curve from time 0 to 12 hours post-dose (AUC0-12) of STP7.
Pharmacokinetics: area under the concentration-time curve from time 0 to 12 hours post-dose of STP7. | Day 10, at pre-dose, 1, 2, 4, 6, 8, 12, 16, 24, 36, and 48 hours post-dose.
  Area under the concentration-time curve from time 0 to 12 hours post-dose (AUC0-12) of STP7.
Pharmacokinetics: area under the concentration-time curve from time 0 to time infinity post-dose of cocaine. | Day 2 and day 10: at 15 minutes before the first infusion, and at 5, 15, 30, 65, 75, 90, 120, 150, and 180 minutes, and at 4, 8, 12, 20 and 32 hours after the first infusion.
  Area under the concentration-time curve from time 0 to time infinity post-dose of cocaine.
Pharmacokinetics: area under the concentration-time curve from time 0 to time infinity post-dose of benzoylecgonine. | Day 2 and day 10: at 15 minutes before the first infusion, and at 5, 15, 30, 65, 75, 90, 120, 150, and 180 minutes, and at 4, 8, 12, 20 and 32 hours after the first infusion.
  Area under the concentration-time curve from time 0 to time infinity post-dose of benzoylecgonine.
Pharmacokinetics: area under the concentration-time curve from time 0 to time infinity post-dose of STP7. | Day 5, day 6, day 7, day 8 and day 9: prior to the morning dose and 4 hours post-dose for each day.
  Area under the concentration-time curve from time 0 to time infinity post-dose of STP7.
Pharmacokinetics: area under the concentration-time curve from time 0 to time infinity post-dose of STP7. | Day 10, at pre-dose, 1, 2, 4, 6, 8, 12, 16, 24, 36, and 48 hours post-dose.
  Area under the concentration-time curve from time 0 to time infinity post-dose of STP7.
Pharmacokinetics: trough plasma concentration (Ctrough) of cocaine. | Day 2 and day 10: at 15 minutes before the first infusion, and at 5, 15, 30, 65, 75, 90, 120, 150, and 180 minutes, and at 4, 8, 12, 20 and 32 hours after the first infusion.
  Trough plasma concentration (Ctrough) of cocaine.
Pharmacokinetics: trough plasma concentration (Ctrough) of benzoylecgonine. | Day 2 and day 10: at 15 minutes before the first infusion, and at 5, 15, 30, 65, 75, 90, 120, 150, and 180 minutes, and at 4, 8, 12, 20 and 32 hours after the first infusion.
  Trough plasma concentration (Ctrough) of benzoylecgonine.
Pharmacokinetics: trough plasma concentration (Ctrough) of STP7. | Day 5, day 6, day 7, day 8 and day 9: prior to the morning dose and 4 hours post-dose for each day.
  Trough plasma concentration (Ctrough) of STP7.
Pharmacokinetics: trough plasma concentration (Ctrough) of STP7. | Day 10, at pre-dose, 1, 2, 4, 6, 8, 12, 16, 24, 36, and 48 hours post-dose.
  Trough plasma concentration (Ctrough) of STP7.
Pharmacokinetics: terminal rate constant of cocaine. | Day 2 and day 10: at 15 minutes before the first infusion, and at 5, 15, 30, 65, 75, 90, 120, 150, and 180 minutes, and at 4, 8, 12, 20 and 32 hours after the first infusion.
  Terminal rate constant of cocaine.
Pharmacokinetics: terminal rate constant of benzoylecgonine. | Day 2 and day 10: at 15 minutes before the first infusion, and at 5, 15, 30, 65, 75, 90, 120, 150, and 180 minutes, and at 4, 8, 12, 20 and 32 hours after the first infusion.
  Terminal rate constant of benzoylecgonine.
Pharmacokinetics: terminal rate constant of STP7. | Day 5, day 6, day 7, day 8 and day 9: prior to the morning dose and 4 hours post-dose for each day.
  Terminal rate constant of STP7.
Pharmacokinetics: terminal rate constant of STP7. | Day 10, at pre-dose, 1, 2, 4, 6, 8, 12, 16, 24, 36, and 48 hours post-dose.
  Terminal rate constant of STP7.
Pharmacokinetics: half-life of cocaine. | Day 2 and day 10: at 15 minutes before the first infusion, and at 5, 15, 30, 65, 75, 90, 120, 150, and 180 minutes, and at 4, 8, 12, 20 and 32 hours after the first infusion.
  Half-life (t1/2) of cocaine
Pharmacokinetics: half-life of benzoylecgonine. | Day 2 and day 10: at 15 minutes before the first infusion, and at 5, 15, 30, 65, 75, 90, 120, 150, and 180 minutes, and at 4, 8, 12, 20 and 32 hours after the first infusion.
  Half-life (t1/2) of benzoylecgonine.
Pharmacokinetics: half-life of STP7. | Day 5, day 6, day 7, day 8 and day 9: prior to the morning dose and 4 hours post-dose for each day.
  Half-life (t1/2) of STP7.
Pharmacokinetics: half-life of STP7. | Day 10, at pre-dose, 1, 2, 4, 6, 8, 12, 16, 24, 36, and 48 hours post-dose.
  Half-life (t1/2) of STP7.
Pharmacokinetics: clearance of cocaine. | Day 2 and day 10: at 15 minutes before the first infusion, and at 5, 15, 30, 65, 75, 90, 120, 150, and 180 minutes, and at 4, 8, 12, 20 and 32 hours after the first infusion.
  Clearance (CL) of cocaine.
Pharmacokinetics: clearance of benzoylecgonine. | Day 2 and day 10: at 15 minutes before the first infusion, and at 5, 15, 30, 65, 75, 90, 120, 150, and 180 minutes, and at 4, 8, 12, 20 and 32 hours after the first infusion.
  Clearance (CL) of benzoylecgonine.
Pharmacokinetics: clearance of STP7. | Day 5, day 6, day 7, day 8 and day 9: prior to the morning dose and 4 hours post-dose for each day.
  Clearance (CL) of STP7.
Pharmacokinetics: clearance of STP7. | Day 10, at pre-dose, 1, 2, 4, 6, 8, 12, 16, 24, 36, and 48 hours post-dose.
  Clearance (CL) of STP7.
Pharmacokinetics: Clearance from plasma after oral administration of cocaine. | Day 2 and day 10: at 15 minutes before the first infusion, and at 5, 15, 30, 65, 75, 90, 120, 150, and 180 minutes, and at 4, 8, 12, 20 and 32 hours after the first infusion.
  Clearance from plasma after oral administration (CL/F) of cocaine.
Pharmacokinetics: Clearance of benzoylecgonine from plasma after oral administration (CL/F) of cocaine. | Day 2 and day 10: at 15 minutes before the first infusion, and at 5, 15, 30, 65, 75, 90, 120, 150, and 180 minutes, and at 4, 8, 12, 20 and 32 hours after the first infusion.
  Clearance of benzoylecgonine from plasma after oral administration (CL/F) of cocaine.
Pharmacokinetics: Clearance from plasma after oral administration (CL/F) of STP7. | Day 5, day 6, day 7, day 8 and day 9: prior to the morning dose and 4 hours post-dose for each day.
  Clearance from plasma after oral administration (CL/F) of STP7.
Pharmacokinetics: Clearance from plasma after oral administration (CL/F) of STP7. | Day 10, at pre-dose, 1, 2, 4, 6, 8, 12, 16, 24, 36, and 48 hours post-dose.
  Clearance from plasma after oral administration (CL/F) of STP7.
Visual evaluation of the STP7 on the subjective effects of cocaine at screening | Day -2: 30 minutes prior to cocaine infusion and at 5, 10, 15, 30, 45, 55, 65, 70, 75, 90, 105, 115, 125, 130, 135, 150, 165 and 180 minutes after the first infusion.
  To evaluate whether STP7 treatment alters the subjective effects of cocaine measured by Visual Analog Scales (VAS).
Visual evaluation of the STP7 on the subjective effects of cocaine at baseline and during treatment | Day 1, day 2, day 9 and day 10: at -30, 5, 10, 15, 30, 45, 55, 65, 70, 75, 90, 105 and 120 minutes after the first infusion.
  To evaluate whether STP7 treatment alters the subjective effects of cocaine measured by Visual Analog Scales (VAS).
Craving evaluation of the STP7 on the subjective effects of cocaine. | Day -2, day 1, day 2, day 9 and day 10: at pre-infusion and 125 minutes after the start of the cocaine infusion.
  To evaluate whether STP7 treatment alters the subjective effects of cocaine on craving measured by the score of the Brief Substance Craving Scale (BSCS).

CONTACTS AND LOCATIONS:
Overall Officials: Debra Kelsh, MD, Principal Investigator — Altasciences Clinical Kansas, Inc.
Locations (1):
- Altasciences Clinical Kansas, Overland Park, Kansas, United States